CLINICAL TRIAL: NCT06035965
Title: Comparison of Quality of Life and Changes Experienced by Patients After Epilepsy Surgery, With Long-term Epileptological Objective Results
Brief Title: Comparison of Quality of Life and Changes Experienced by Patients After Epilepsy Surgery
Acronym: EPICHANGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0411
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Epilepsy Surgery Satisfaction Questionnaire (ESSQ-19) — 19 items assessing post-surgery satisfaction.
Other: Quality of Life in Epilepsy Inventory (QOLIE-31) — 31 items to assess different dimensions of quality of life
Other: Generalized Anxiety Disorder 7 (GAD7) — 7 items, rated from 0 to 3, to detect anxiety disorders.
Other: Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) — to screen for depressive disorders
Other: Evaluation of Changes in Daily Life after Epilepsy Surgery (EVOCQUE) — self-questionnaire developed by the Toulouse epileptology team in 2023 for patients who have undergone epilepsy surgery. It aims to collect the feelings of patients concerning the changes induced by surgery in their daily life according to a 7-point Likert scale.

SUMMARY:
Epilepsy is one of the most common chronic neurological diseases. According to data from the World Health Organization (WHO), it affects 0.5 to 1% of the population, or around 70 million people world-wide and around 600,000 in France. There are several more or less severe forms of epilepsy depending on the type of epileptic seizures and the frequency of these seizures. About 30% of epileptic patients respond poorly to well-conducted medical treatment, which makes the number of so-called "drug-resistant" patients estimated at between 100,000 and 150,000 patients.

Epilepsy surgery is possible in some cases of drug-resistant epilepsy and can lead to complete seizure control. Beyond the impact on the control of seizures, surgery can have an impact on the lives of patients at the psychological, emotional and cognitive level, with consequences on their socio-professional but also personal life. Thus the impact on the daily life of patients after epilepsy surgery can vary greatly from one patient to another and the personal feelings of operated patients do not always seem to correspond to the objective elements collected by doctors. 2.3 The investigators want to retrospectively assess the satisfaction and quality of life of patients operated on for more than 2 years based on their epileptological results (frequency of seizures).

ELIGIBILITY:
Inclusion Criteria:

* Patient operated in the context of epilepsy surgery dating back more than 2 years in the epileptology center of the Toulouse University Hospital.
* Patient covered by a social security scheme.
* Patient having given his non-objection to participate in the research.

Exclusion Criteria:

* Minor under the age of 15 at the time of the questionnaires.
* Serious psychiatric pathology unrelated to epilepsy surgery.
* Severe intellectual disability limiting responses to self-questionnaires.
* Language barrier.
* Patients under guardianship and protection of justice.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient operated in the context of epilepsy surgery dating back more than 2 years in the epileptology center of the Toulouse University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the changes felt by patients | 2 years
  Evaluate the changes felt by patients more than 2 years after surgery in the context of drug-resistant epilepsy using a new questionnaire created by the epileptology team of the Toulouse University Hospital. The rating of the responses is distributed between 0 and 100 (0 = very negative change, 50 = no change and 100 = very positive change).

CONTACTS AND LOCATIONS:
Overall Officials: HELENE MIRABEL, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No